CLINICAL TRIAL: NCT01290354
Title: An Open-label Positron Emission Tomography Study to Investigate and Quantify Brain and Tumour Penetration of [11C]Lapatinib in Subjects With HER2-overexpressing Breast Cancer
Brief Title: Exploratory Lapatinib (Positron Emission Tomography) PET Study in Subjects With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 112867
Record Dates: First submitted 2011-01-27; First posted 2011-02-07 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: Brain penetration; positron emission tomography; Lapatinib
MeSH Terms: conditions — Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lapatinib (Experimental): unlabelled, administered orally
  Interventions: Drug: Lapatinib; Drug: [11C] lapatinib

INTERVENTIONS:
Drug: Lapatinib — Unlabelled, administered orally
  Other Names: Tykerb; Tyverb
Drug: [11C] lapatinib — Radiolabelled, administered intravenously

SUMMARY:
The purpose of this study is to find out how much lapatinib can enter both normal brains and brains in which tumours secondary to breast cancer have developed.

DETAILED DESCRIPTION:
Lapatinib is an anti-cancer drug taken by mouth which inhibits the HER2 protein, overexpressed in some breast tumours. It is not known whether lapatinib passes through the blood-brain barrier, and, therefore, whether it can target secondary tumours in the brain. This study will investigate whether lapatinib does indeed enter the brain.

Subjects with HER2-overexpressing breast cancer, with and without brain metastases, will receive lapatinib tablets daily for 8 days. The subjects will also receive lapatinib with a small amount of radioactivity attached on the first and last days of dosing to investigate whether it is taken up by the brain, using positron emission tomography (PET) scans.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged >/= 18 years old
* Advanced or metastatic breast cancer with overexpression of HER2
* Be able to provide written informed consent and comply with protocol requirements
* If of child-bearing potential, using adequate and medically acceptable contraception method
* Have an ECOG performance status of 0-2 and be in stable condition
* Able to lie still on the PET scanner for approx. 1.5-2 h
* Adequate hepatic and renal function
* Patent ulnar artery or collateral arterial blood vessels
* If have CNS metastases, disease must be stable
* Subjects with CNS metastases should have at least a single 1 cm diameter lesion as shown on contrast MRI

Exclusion Criteria:

* Subjects with brain metastases who have undergone prior CNS surgery
* Significant brain abnormalities, neurological disorder, psychiatric disorder or previous brain damage
* Diabetes type I
* History of HIV, hepatitis B or hepatitis C infection
* Current alcohol and/or drug abuse
* Positive pregnancy test or lactation
* Malabsorption syndrome or disease affecting gastrointestinal function that may affect intestinal absorption
* Requirement for additional concurrent anti-cancer therapy
* History of uncontrolled or symptomatic angina
* Concurrent treatment with an investigational agent or anti-cytotoxic therapy or use within 30 days or 5 half-lives
* Known hypersensitivity reaction of idiosyncrasy to drugs chemically related to lapatinib or its excipients
* Concurrent treatment with CYP3A4 inducers and inhibitors
* Unwillingness to refrain from consuming red wine, Seville oranges, grapefruit, pomelo, grapefruit hybrids and their juices from 7 days before Day 1 until collection of the final pharmacokinetic sample
* Known history of claustrophobia
* Known contraindications or likely risk of toxicity to gadlinium-based MRI contrast media
* Presence of cardiac pacemaker, other electronic device or ferromagnetic metal foreign bodies
* Any abnormality found on the MRI scan which, in the opinion of the investigator, may influence the outcome of the PET scans or affect the safety of the volunteer
* Acute or active hepatic or biliary disease
* Any medical condition or circumstance making the volunteer unsuitable for participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2013-03-18 (Actual)

PRIMARY OUTCOMES:
Brain penetration of [11C]lapatinib | 8 days
Brain tumour penetration of [11C]lapatinib | 8 days

SECONDARY OUTCOMES:
Safety as assessed by number of subjects with adverse events | 16-19 days
[11C]lapatinib uptake in non-brain tumour sites | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Saleem A, Searle GE, Kenny LM, Huiban M, Kozlowski K, Waldman AD, Woodley L, Palmieri C, Lowdell C, Kaneko T, Murphy PS, Lau MR, Aboagye EO, Coombes RC. Lapatinib access into normal brain and brain metastases in patients with Her-2 overexpressing breast cancer. EJNMMI Res. 2015 Apr 30;5:30. doi: 10.1186/s13550-015-0103-5. eCollection 2015. PMID 25977884
- See also: Results for study 112867 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112867?search=study&study_ids=112867#rs